CLINICAL TRIAL: NCT04635449
Title: A Prospective Randomised Controlled Study of a Directed Psycho-educational Tool to Prevent Psychological Sequelae Following Paediatric Intensive Care Admission.
Brief Title: Psycho-educational Tool to Prevent Psychological Sequelae Following Paediatric Intensive Care Unit Admission
Acronym: 4PICU
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20SM6281
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group, single centre, randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): age-specific information, complemented by a follow-up targeted telephone call
  Interventions: Other: Age-specific information booklet and targeted telephone call
- Treatment as usual (No Intervention): usual information given at PICU discharge

INTERVENTIONS:
Other: Age-specific information booklet and targeted telephone call — age-specific information, complemented by a follow-up targeted telephone call to reduce psychological sequelae in the child and their parents after PICU discharge.
  Arms: Intervention

SUMMARY:
* To systematically evaluate an innovative directed psycho-educational intervention consisting of written specific, age-appropriate information, complemented by a follow-up targeted telephone call in order to reduce psychological sequelae in the child and their parents/guardians after PICU discharge.
* To confirm the effects of the psycho-educational tool on parent and child emotional adjustment 6 months after PICU discharge; and to explore whether these outcomes are associated with the child's age; with receipt of the targeted telephone call; and/or with parental levels of stress during the child's admission.
* To obtain detailed feedback from parents/guardians and children about the different aspects of the psycho-educational intervention (the written information and the targeted telephone call) and the utility of these two psycho-educational interventions.

The study team will perform a randomised controlled trial of the intervention vs treatment as usual in children 0-16 years, stratified according to age (< 4 years and > 4 years).

It is estimated that 288 children will be required to show a difference in outcome which is PTSD in parents and children.

DETAILED DESCRIPTION:
STUDY OBJECTIVES AND PURPOSE

Aims

* To systematically evaluate an innovative directed psycho-educational intervention consisting of written specific, age-appropriate information, complemented by a follow-up targeted telephone call in order to reduce psychological sequelae in the child and their parents/guardians after PICU discharge.
* To confirm the effects of the psycho-educational tool on parent and child emotional adjustment 6 months after PICU discharge; and to explore whether these outcomes are associated with the child's age; with receipt of the targeted telephone call; and/or with parental levels of stress during the child's admission.
* To obtain detailed feedback from parents/guardians and children about the different aspects of the psycho-educational intervention (the written information and the targeted telephone call) and the utility of these two psycho-educational interventions.

Primary Objective To determine if the psycho-educational intervention is superior to treatment as usual in reducing parental post-traumatic stress and other psychological symptoms measured at 6 months after PICU discharge.

Secondary Objectives

* To determine if the intervention is superior to treatment as usual in reducing child post-traumatic stress and other psychological symptoms measured at 6 months post PICU discharge.
* To determine whether the degree of parental stress during their child's PICU admission is particularly associated with the extent of psychological sequelae and whether the psycho-educational intervention is as less or more effective in the highly stressed families.
* To determine if adding this relatively simple, innovative and pragmatic intervention to treatment as usual will provide a cost-effective use of NHS resources
* To evaluate in detail child and parental acceptance of the intervention.

Delivery of the Psycho-educational Tool and Assessment of Parental/Guardian Stress on PICU Discharge

* Eligible families will include children 0-16 years admitted to PICU for > 24 hours, surviving to be discharged.
* Parents who are deemed to lack adequate English Language to understand the written psycho-educational tool, telephone call and questionnaires will be excluded.

[Our aim in future, if the intervention is shown to be successful, is to translate the intervention tools into the most frequently encountered foreign languages.]

After obtaining informed consent prior to the child's discharge from PICU, a parental PICU stress screening questionnaire (18), will be given to all parents/guardians prior to discharge by the researcher or appropriately trained bedside PICU nurse.

* Parents/guardians of all eligible children will be randomized using random allocation to receive either active intervention or treatment as usual (TAU).
* Those randomised to the intervention group will be given the age-appropriate written psycho-educational tool prior to PICU discharge, by the researcher. The researcher will also explain the mechanism of the targeted telephone call to be delivered 4-6 weeks after PICU discharge.

  • Telephone Call:
* All parents/guardians randomised to the intervention group will be offered the directed targeted telephone call from the researcher at 4-6 weeks post hospital discharge.
* The researcher will use a protocolised, scripted interview questionnaire to discuss the contents of the tool and any psychological problems arising post PICU discharge, as well as provide information to families of ways of managing these, including, when appropriate referral to GP and local mental health services.
* The study team will record the key outcomes of the call to include:

Uptake rates and outcome; the number of families with impairing symptoms; and rates of referral to GPs and/or local mental health services.

ELIGIBILITY:
Inclusion Criteria:

* All children and young people age 0-16 years
* > 36 weeks corrected gestational age
* Admitted to PICU >24 hours Parent(s)/guardian aged >18 years

Exclusion Criteria:

* • Children where treatment withdrawal is being considered

  * Life expectancy <6 months
  * Previous admission to Paediatric, or Neonatal Intensive Care for > 24 hours, in the last 12months preceding the current PICU admission
  * Parent(s)/ guardian to have insufficient English to complete questionnaires
  * Overseas address

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 288 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
post-traumatic stress symptoms in the parents/guardians | 6 months post PICU discharge
  measured using the Impact of Events Scale, a self-report questionnaire

SECONDARY OUTCOMES:
Parent/guardian general emotional state | 6 months post PICU discharge
  Hospital Anxiety and Depression Questionnaire
Child post-traumatic stress and other emotional and behavioural problems | 6 months post PICU discharge
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Simon Nadel, MBBS, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Will share will other researchers within Imperial

REFERENCES:
- [Derived] Bridges K, Vickers B, Mitting RB, Cooper M, Garralda E, Nadel S. Directed psychoeducational tool to prevent psychological sequelae following paediatric intensive care admission: a prospective randomised controlled study (the 4PICU study). Arch Dis Child. 2026 Jan 19;111(2):133-140. doi: 10.1136/archdischild-2025-328691. PMID 41015488